CLINICAL TRIAL: NCT03724292
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VTP-43742 in Healthy Volunteers and Proof-of-Concept in Psoriatic Patients
Brief Title: An Ascending Multiple Dose Study With VTP-43742 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vitae Pharmaceuticals Inc., an Allergan affiliate (Industry)
Responsible Party: Sponsor
Organization: Vitae Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VTP-43742-002-1
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Psoriasis
Keywords: Moderate to severe chronic plaque-type psoriasis
MeSH Terms: conditions — Psoriasis | interventions — VTP-43742

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Dose-matched placebo administered as oral capsule(s) once daily
  Interventions: Drug: Placebo
- VTP-43742 Dose 1 (Experimental): VTP-43742 administered as oral capsule(s) once daily
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 2 (Experimental): VTP-43742 administered as oral capsule(s) once daily
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 3 (Experimental): VTP-43742 administered as oral capsule(s) once daily
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 4 (Experimental): VTP-43742 administered as oral capsule(s) once daily
  Interventions: Drug: VTP-43742
- VTP-43742 Dose 5 (Experimental): VTP-43742 administered as oral capsule(s) once daily
  Interventions: Drug: VTP-43742

INTERVENTIONS:
Drug: Placebo — Dose-matched placebo administered as oral capsule(s) once daily
  Arms: Placebo
Drug: VTP-43742 — VTP-43742 administered as oral capsule(s) once daily
  Arms: VTP-43742 Dose 1; VTP-43742 Dose 2; VTP-43742 Dose 3; VTP-43742 Dose 4; VTP-43742 Dose 5

SUMMARY:
This is Part 1 of a two-part, randomized, double-blind, placebo-controlled study in which VTP-43742 was administered to participants; Part 1 in healthy volunteers and Part 2 in psoriatic participants.

DETAILED DESCRIPTION:
This was a prospective, randomized, double-blind, placebo-controlled, ascending multiple dose study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics effects of VTP-43742 in healthy volunteers conducted at a single, study center in the United States (Part 1). A total of 74 participants were enrolled both parts of the study (Part 1 with 40 healthy subjects; Part 2 with 34 psoriatic participants). This post includes data from Part 1 of the study only; Part 2 is reported separately.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, 18 to 45 years of age, inclusive.
* Body weight of at least 55 kg and body mass index of 18-32 kg/m2, inclusive.
* Medically healthy with clinically insignificant screening results.
* Women of child-bearing potential (WOCBP) AND men with partners who are WOCBP must agree that they and/or their partner will use two reliable forms of contraception as per study requirements
* WOCBP must have a negative serum β-hCG pregnancy test at the Screening and Baseline visit.
* Voluntarily consent to participate in the trial

Exclusion Criteria:

* Unwilling or unable to provide written informed consent
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, coagulation, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Evidence of organ dysfunction or any clinically significant deviation from normal in vital signs, physical examination, clinical laboratory determinations or ECG
* Any major surgery within 3 months of Screening
* Positive urine drug/alcohol testing at Screening or Baseline visit
* Use of tobacco and/or nicotine-containing products within 3 months prior to the start of dosing of the trial
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV Ab) at Screening
* History or presence of alcoholism or drug abuse as defined in DSM V, Diagnostic Criteria for Drug and Alcohol Abuse
* History of hypersensitivity or idiosyncratic reaction to drugs from multiple drug classes
* Any previous gastrointestinal surgery or recent (within 3 months) history of gastrointestinal disease that could impact the absorption of the study drug
* Blood donation or significant blood loss within 8 weeks prior to Day 1 of the trial
* Plasma donation within 7 days prior to Day 1 of the trial
* Blood transfusion within 4 weeks of Screening
* Positive serum pregnancy test (WOCBP) at the Screening or Baseline visit
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical disease (e.g., infectious disease) must not be enrolled into this study
* Any other medical, psychiatric, and/or social reason as determined by the Investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-03-08 (Actual); Study Completion 2016-03-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) in the healthy volunteer (Part 1) group | Study Day 1 to Day 17±2 (follow up)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) in the healthy volunteer (Part 1) group | Day 1 and Day 10
Time to maximum plasma concentrations (tmax) in the healthy volunteer (Part 1) group | Day 1 and Day 10
The area under the plasma concentration versus time curve, from time 0 to the last measurable concentration (AUCt) in the healthy volunteer (Part 1) group | Day 1 and Day 10
Half life (t½) in the healthy volunteer (Part 1) group | Day 10 to Day 13 (72 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gregg, MD, Study Director — Vitae Pharmaceuticals
Locations (1):
- Healthy Volunteer Site 1, Fair Lawn, New Jersey, United States